CLINICAL TRIAL: NCT04507880
Title: A 2-Year Prospective Follow-up Study of the Global Unite Reverse Fracture Shoulder System for Proximal Humerus Fractures
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Signe Rosner Rasmussen (Other)
Collaborators: Herlev and Gentofte Hospital (Other)
Responsible Party: Sponsor-Investigator, Signe Rosner Rasmussen, MD, orthopedic resident, principal investigator, Herlev and Gentofte Hospital
Organization: Herlev and Gentofte Hospital (Other)
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 71005
Record Dates: First submitted 2020-07-31; First posted 2020-08-11 (Actual); Last update posted 2020-08-11 (Actual); Status verified 2020-07

CONDITIONS: Shoulder Fractures
Keywords: Humeral Fractures, Proximal
MeSH Terms: conditions — Shoulder Fractures | interventions — Hemiarthroplasty

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- RTSA group (Experimental): Participants with a complex proximal humerus fracture given a RTSA
  Interventions: Device: Reverse Total Shoulder Arthroplasty
- Hemiarthroplasty group (Active Comparator): Historical cohort of participants, operated with a hemiarthroplasty of the shoulder
  Interventions: Device: Hemiarthroplasty

INTERVENTIONS:
Device: Reverse Total Shoulder Arthroplasty — The RTSA (GLOBAL UNITE Reverse Fracture System) from DePuy Synthes.
  Arms: RTSA group
Device: Hemiarthroplasty — The shoulder hemiarthroplasty
  Arms: Hemiarthroplasty group

SUMMARY:
The objective of this study is to evaluated the efficacy and safety of the reverse total shoulder prosthesis (RTSA) for complex proximal humerus fractures. The clinical results of RTSA will be compared to clinical results from a historical cohort, that received a hemiarthroplasty of the shoulder.

ELIGIBILITY:
Inclusion Criteria:

* Fracture or fracture dislocation not suitable for non-operative treatment or for osteosynthesis due to displacement and comminution
* Patients older than 65-years of age, or younger than 65-year of age if the surgeon assesses the physiological age as older.
* All patients, regardless of age, with an insufficient or irreparable rotator cuff

Exclusion Criteria:

* Brachial plexus palsy
* Previous ipsilateral fracture of clavicula, scapula, or proximal humerus
* Cognitive disabilities or substance abuse enabling rehabilitation and follow-up
* Patients without a Danish civil registration number

Ages: 65 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2020-08-01 (Estimated); Primary Completion 2024-08-01 (Estimated); Study Completion 2024-08-01 (Estimated)

PRIMARY OUTCOMES:
Change in Constant score (CS) | The outcome is measured 3 months, 6 months, 1 year and 2 years after surgery
  The CS consists of four parameters (pain, mobility, ADL, strength) assessing shoulder function after the treatment of shoulder injury, both subjectively and objectively. The scale rates from worst (0) to best (100) quality of shoulder function.

SECONDARY OUTCOMES:
Change in Oxford Shoulder Score (OSS) | The outcome is measured 3 months, 6 months, 1 year and 2 years after surgery
  The OSS is a patient related outcome-measure (PROM) validated for evaluating self-assessed functionality after shoulder surgery. The 12 questions, with five response options, gives a total score ranging from 12 points (no pain or functional impairment) to 60 points (worst).
Change in Western Ontario Osteoarthritis of the Shoulder Index (WOOS) | The outcome is measured 3 months, 6 months, 1 year and 2 years after surgery
  The WOOS is a patient-related outcome measurement, initially validated for patients with osteoarthritis of the shoulder. On four domains (physical symptoms, recreation/work, lifestyle, emotions) the visual analog scale measures shoulder-related quality-of-life with a maximum of 1900 points, which signifies highest quality of function.
Change in EQ5D questionnaire | The outcome is measured 3 months, 6 months, 1 year and 2 years after surgery
  The EQ-5D (EuroQuol 5 Dimension scale) questionnaire is a widely used patient-related outcome measurement for quality of life assessment in general, consisting of 25 dichotomous questions from five parameters and a visual analog scale to plot perceived health. A persons selfperceived health status is then evaluated as a 5-digit number, ranging from 11111 (having no problems) to 33333 (having problems in all 5 aspects), and as a number from 0 (worst imaginable health) to 100 (best imaginable health).
Change in Numeric Ranking Scale | The outcome is measured 3 months, 6 months, 1 year and 2 years after surgery
  Pain measured after surgery according to the Numeric Ranking Scale (NRS), where 0 is no pain and 10 is worst imaginable pain.
Complications | The outcome is registered 2 years after surgery
  Postoperative complications or reoperation due to infection, nerve damage, vascular damage, iatrogenic perioperative fracture, or loosening of the implant.
Change in humeral tuberosities | The outcome is measured 3 months, 6 months, 1 year and 2 years after surgery
  Migration or resorption of the humeral tuberosities accessed qualitatively from the xrays.

CONTACTS AND LOCATIONS:
Overall Officials: Bo S Olsen, Professor, Study Chair — Herlev and Gentofte Hospital

IPD SHARING:
Plan to Share IPD: No